CLINICAL TRIAL: NCT03140488
Title: High Dose vs. Low Dose Oxytocin for Labor Induction in Obese Women: a Randomized Controlled Trial - the OPS (Obese Pitocin Study) Trial
Brief Title: Oxytocin Dosage to Decrease Induction Duration
Acronym: OPS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, Meghan Hill, Assistant Professor, University of Arizona
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 1702231223
Record Dates: First submitted 2017-04-19; First posted 2017-05-04 (Actual); Results first posted 2022-12-20 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-11

CONDITIONS: Obesity; Labor, Induced; Oxytocin
Keywords: Induction of labor; Pitocin; BMI
MeSH Terms: conditions — Obesity | interventions — Oxytocin

STUDY DESIGN:
Intervention Model Description: 4 Comparison groups:
  1. Control group: Lean cohort: BMI ≤25, at <20 weeks gestation or BMI ≤28 at a term gestation, low dose oxytocin protocol
  2. Intervention group: Lean cohort: BMI ≤25, at <20 weeks gestation or BMI ≤28 at a term gestation, high dose oxytocin protocol
  3. Control group: Obese cohort: BMI ≥30, at <20 weeks gestation or BMI ≥35 at a term gestation, low dose oxytocin protocol
  4. Intervention group: Obese cohort: BMI ≥30, at <20 weeks gestation or BMI ≥35 at a term gestation, high dose oxytocin protocol
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This portion of the study will be carried out by the research pharmacy. Single (low dose) and triple (high dose) concentration of oxytocin will be premixed in the intravenous fluid bag in the pharmacy. Sequence generation for randomization will be created with 1:1 ratio in both the obese and lean group by the Department of Statistics. After the sequence is generated, ths list will be given to the research pharmacy. The premixed oxytocin medication will be sequentially labelled as "OPS drug, patient #1, 2, 3" etc. per the allocation. Allocation concealment will also be carried out by pharmacy as these bags will completely appear identical after they are labelled numerically. Once a patient is randomized, the pharmacy will send up the appropriate concentration of oxytocin already premixed in the intravenous fluid bag, labelled as "OPS drug, patient #". Lean group will be assigned at # 1-70 and obese group will be assigned at #71-140.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Lean-Control (Active Comparator): 1) Control group: Lean cohort: BMI ≤25, at <20 weeks gestation or BMI ≤28 at a term gestation, low dose oxytocin protocol
  Low dose oxytocin regimen (the standard at Banner University Labor and Delivery, as well as across the United States): 30 units in 500cc 0.9% normal saline bag (60 milliunit/cc). Starting rate would be 2 milliunit/minute, or 2cc/hour. The medication will be increased by 2 milliunit/minute = 2cc/hr every 30 minutes until adequacy of contraction or cervical change. At 20 milliunit/minute = 20cc/hr, provider will assess patient for eligibility to continue to increase oxytocin dosage.
  Interventions: Drug: Oxytocin
- Lean-Intervention (Experimental): 2) Intervention group: Lean cohort: BMI ≤25, at <20 weeks gestation or BMI ≤28 at a term gestation, high dose oxytocin protocol
  High dose oxytocin regimen (endorsed by American College of Obstetricians and Gynecologists): 90 units in 500cc 0.9% normal saline bag (180 milliunit/cc). Starting rate would be 6 milliunit/minute, or 2cc/hour. The medication will be increased by 6 milliunit/minute = 2cc/hr every 30 minutes until adequacy of contraction or cervical change. At 60 milliunit/minute = 20cc/hr, provider will assess patient for eligibility to continue to increase oxytocin dosage.
  Interventions: Drug: Oxytocin
- Obese-Control (Active Comparator): 3) Control group: Obese cohort: BMI ≥30, at <20 weeks gestation or BMI ≥35 at a term gestation, low dose oxytocin protocol
  Low dose oxytocin regimen (the standard at Banner University Labor and Delivery, as well as across the United States): 30 units in 500cc 0.9% normal saline bag (60 milliunit/cc). Starting rate would be 2 milliunit/minute, or 2cc/hour. The medication will be increased by 2 milliunit/minute = 2cc/hr every 30 minutes until adequacy of contraction or cervical change. At 20 milliunit/minute = 20cc/hr, provider will assess patient for eligibility to continue to increase oxytocin dosage.
  Interventions: Drug: Oxytocin
- Obese-Intervention (Experimental): 4) Intervention group: Obese cohort: BMI ≥30, at <20 weeks gestation or BMI ≥35 at a term gestation, high dose oxytocin protocol
  High dose oxytocin regimen (endorsed by American College of Obstetricians and Gynecologists): 90 units in 500cc 0.9% normal saline bag (180 milliunit/cc). Starting rate would be 6 milliunit/minute, or 2cc/hour. The medication will be increased by 6 milliunit/minute = 2cc/hr every 30 minutes until adequacy of contraction or cervical change. At 60 milliunit/minute = 20cc/hr, provider will assess patient for eligibility to continue to increase oxytocin dosage.
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Oxytocin — Patients will be randomized to low dose or high dose oxytocin for induction of labor.
  Other Names: Pitocin; Syntocinon

SUMMARY:
This is a randomized controlled trial in which women are allocated either 'high dose' or 'low dose' oxytocin infusions for induction of labour. The randomization is stratified by maternal body mass index.

DETAILED DESCRIPTION:
Obesity is considered a major public health concerns and increases the risk of many comorbid medical conditions. Obesity in pregnancy places women at higher risk of obstetrical complications during pregnancy, delivery and postpartum. In particular, obese pregnant women have more difficulty going into labor, a longer labor course, and even with pharmacologic treatment, have a higher chance of requiring cesarean delivery.

When pregnant women need help going into labor, they commonly receive a medication called Pitocin on the labor and delivery floor. Pitocin is the brand name and is a synthetic analog to the naturally produced oxytocin, a hormone secreted by mother when they naturally go into labor. This medication has been used widely around the world. There is emerging evidence that obese women need more oxytocin to go into labor compared to their lean cohorts. There are many studies to support the use of different oxytocin dosage protocols (both high and low dose infusion increments). Despite these evidences, a low dose oxytocin regimen is universally used in the United States, regardless of patient characteristics.

This study is a double blinded randomized controlled trial. Both lean and obese cohorts will be recruited for the study. The investigators will randomly place both cohorts into the low or the high dose oxytocin regimen treatment group. The investigators, patients and providers will be blinded and will not know the specific assignments. The purpose of this study is to evaluate the effect of high dose oxytocin in the obese cohort. The hypothesis is that obese patient will have shorter time to delivery with the high dose oxytocin regimen without incurring any additional risks or adverse outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy ≥ 37 weeks gestation
* Patient presented for induction of labor who is determined to be a candidate for oxytocin
* Cephalic presentation
* Reassuring fetal health assessment (no abnormal findings in fetal assessment, see below)
* Meeting one of the following BMI category:

Obese group: BMI ≥30 at <20 weeks of pregnancy, or BMI ≥35 at a term gestation of pregnancy Lean group: BMI ≤25 at <20 weeks of pregnancy, or BMI ≤28 at a term gestation of pregnancy

Exclusion Criteria:

* Non-reassuring fetal assessment at the time of recruitment
* Previous cervical ripening agents (cytotec, cervidil, cervical Foley Balloon)
* <18 years of age
* Prisoners
* Any patients contraindicated for vaginal delivery
* Multiple gestations
* History of previous cesarean delivery
* Patients with history of significant cardiac disease
* Fetal demise
* Estimated fetal weight greater than 4500 grams in diabetic and 5000 grams in non-diabetic mother
* Ruptured membranes
* Spontaneous labor (latent or active phase)
* Augmentation of labor (latent or active phase)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2017-06-05 (Actual); Primary Completion 2018-10-12 (Actual); Study Completion 2019-09-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Meghan Hill, MBBS, Principal Investigator — University of Arizona
Locations (1):
- Banner University Medical Center Tucson, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wei RM, Bounthavong M, Hill MG. High- vs low-dose oxytocin in lean and obese women: a double-blinded randomized controlled trial. Am J Obstet Gynecol MFM. 2022 Jul;4(4):100627. doi: 10.1016/j.ajogmf.2022.100627. Epub 2022 Mar 28. PMID 35358738

RESULTS

PARTICIPANT FLOW:
Groups:
- Lean-Intervention: 2) Intervention group: Lean cohort: BMI ≤25, at <20 weeks gestation or BMI ≤28 at a term gestation, high dose oxytocin protocol
  High dose oxytocin regimen (endorsed by American College of Obstetricians and Gynecologists): 90 units in 500cc 0.9% normal saline bag (180 milliunit/cc). Starting rate would be 6 milliunit/minute, or 2cc/hour. The medication will be increased by 6 milliunit/minute = 2cc/hr every 30 minutes until adequacy of contraction or cervical change. At 60 milliunit/minute = 20cc/hr, provider will assess patient for eligibility to continue to increase oxytocin dosage.
  Oxytocin: Patients will be randomized to low dose or high dose oxytocin for induction of labor.
- Obese-Intervention: 4) Intervention group: Obese cohort: BMI ≥30, at <20 weeks gestation or BMI ≥35 at a term gestation, high dose oxytocin protocol
  High dose oxytocin regimen (endorsed by American College of Obstetricians and Gynecologists): 90 units in 500cc 0.9% normal saline bag (180 milliunit/cc). Starting rate would be 6 milliunit/minute, or 2cc/hour. The medication will be increased by 6 milliunit/minute = 2cc/hr every 30 minutes until adequacy of contraction or cervical change. At 60 milliunit/minute = 20cc/hr, provider will assess patient for eligibility to continue to increase oxytocin dosage.
  Oxytocin: Patients will be randomized to low dose or high dose oxytocin for induction of labor.
Period: Overall Study
Arm/Group | Lean-Control | Lean-Intervention | Obese-Control | Obese-Intervention
Started | 35 | 35 | 35 | 35
Completed | 35 | 35 | 35 | 35
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lean-Control | Lean-Intervention | Obese-Control | Obese-Intervention | Total
Number analyzed (Participants) | 35 | 35 | 35 | 35 | 140
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 35 | 35 | 35 | 35 | 140
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.89 (5.76) | 28.54 (5.2) | 30.63 (5.31) | 26.80 (4.51) | 28.71 (5.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 35 | 35 | 35 | 140
  Male | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 4 | 4 | 1 | 0 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 2 | 2 | 6
  White | 30 | 28 | 32 | 33 | 123
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 0 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 35 | 35 | 35 | 35 | 140

OUTCOME MEASURES:

1. Primary Outcome: Length of Time to Delivery
Description: Number of minutes from induction of labor with oxytocin infusion to delivery of infant, no maximum amount of time specified.
Time Frame: Start of induction to Delivery
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Lean-Control | Lean-Intervention | Obese-Control | Obese-Intervention
Number analyzed (Participants) | 29 | 33 | 30 | 34
minutes | 796 (411) | 694 (466) | 715 (497) | 762 (594)

2. Secondary Outcome: Maximum Oxytocin Infusion Rate
Description: rate measured in milliunits/minute during induction of labour, no time limit applied.
Time Frame: Start of induction to Delivery
Measure: Mean (Standard Deviation); unit: milliunits per minute
Arm/Group | Lean-Control | Lean-Intervention | Obese-Control | Obese-Intervention
Number analyzed (Participants) | 26 | 20 | 22 | 20
milliunits per minute | 14.85 (7.16) | 33.00 (25.64) | 17.14 (10.99) | 39.60 (21.09)

3. Secondary Outcome: Number of Participants With Terbutaline Use
Description: If terbutaline was injected during labor to decrease number or strength of contraction
Time Frame: Start of induction to Delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Lean-Control | Lean-Intervention | Obese-Control | Obese-Intervention
Number analyzed (Participants) | 35 | 35 | 35 | 35
Participants | 0 | 0 | 0 | 1

4. Secondary Outcome: Rate of Cesarean Delivery
Description: total number of patients who undergo cesarean delivery
Time Frame: Start of induction to Delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Lean-Control | Lean-Intervention | Obese-Control | Obese-Intervention
Number analyzed (Participants) | 35 | 35 | 35 | 35
Participants | 5 | 2 | 4 | 1

5. Secondary Outcome: Rate of Cesarean Delivery for Labor Arrest
Description: Number of patients who undergo cesarean delivery due to labor arrest/ failed induction
Time Frame: Start of induction to Delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Lean-Control | Lean-Intervention | Obese-Control | Obese-Intervention
Number analyzed (Participants) | 35 | 35 | 35 | 35
Participants | 1 | 1 | 3 | 0

6. Secondary Outcome: Maternal Blood Loss
Description: Blood loss in milliliters
Time Frame: At delivery
Measure: Mean (Standard Deviation); unit: milliliters
Arm/Group | Lean-Control | Lean-Intervention | Obese-Control | Obese-Intervention
Number analyzed (Participants) | 35 | 35 | 35 | 35
milliliters | 391.14 (207.96) | 358.57 (166.49) | 404.29 (226.99) | 491.43 (342.89)

7. Secondary Outcome: Number of Neonates With Apgar Score <7
Description: 5 minute Apgar Score <7
  *Apgar is an acronym for which each criterion is given a minimum of 0 and maximum of 2 points: Appearance (skin color), Pulse (heart rate), Grimace (reflex irritability), Activity (muscle tone), Respiration
Time Frame: 5 minutes after birth
Measure: Count of Participants; unit: Participants
Arm/Group | Lean-Control | Lean-Intervention | Obese-Control | Obese-Intervention
Number analyzed (Participants) | 35 | 35 | 35 | 35
Participants | 0 | 3 | 0 | 1

ADVERSE EVENTS:
Time Frame: From start of oxytocin infusion until discharge from hospital after birth. We did not specify a number of days after giving birth we would collect adverse event data. However, no participants had data collected past 1 month from giving birth.
Groups:
- Lean-Control: 1) Control group: Lean cohort: BMI ≤25, at <20 weeks gestation or BMI ≤28 at a term gestation, low dose oxytocin protocol
  Low dose oxytocin regimen (the standard at Banner University Labor and Delivery, as well as across the United States): 30 units in 500cc 0.9% normal saline bag (60 milliunit/cc). Starting rate would be 2 milliunit/minute, or 2cc/hour. The medication will be increased by 2 milliunit/minute = 2cc/hr every 30 minutes until adequacy of contraction or cervical change. At 20 milliunit/minute = 20cc/hr, provider will assess patient for eligibility to continue to increase oxytocin dosage.
  Time frame measured from start of oxytocin infusion until the mother is discharged from hospital after giving birth.
- Lean-Intervention: 2) Intervention group: Lean cohort: BMI ≤25, at <20 weeks gestation or BMI ≤28 at a term gestation, high dose oxytocin protocol
  High dose oxytocin regimen (endorsed by American College of Obstetricians and Gynecologists): 90 units in 500cc 0.9% normal saline bag (180 milliunit/cc). Starting rate would be 6 milliunit/minute, or 2cc/hour. The medication will be increased by 6 milliunit/minute = 2cc/hr every 30 minutes until adequacy of contraction or cervical change. At 60 milliunit/minute = 20cc/hr, provider will assess patient for eligibility to continue to increase oxytocin dosage.
  Time frame measured from start of oxytocin infusion until the mother is discharged from hospital after giving birth.
- Obese-Control: 3) Control group: Obese cohort: BMI ≥30, at <20 weeks gestation or BMI ≥35 at a term gestation, low dose oxytocin protocol
  Low dose oxytocin regimen (the standard at Banner University Labor and Delivery, as well as across the United States): 30 units in 500cc 0.9% normal saline bag (60 milliunit/cc). Starting rate would be 2 milliunit/minute, or 2cc/hour. The medication will be increased by 2 milliunit/minute = 2cc/hr every 30 minutes until adequacy of contraction or cervical change. At 20 milliunit/minute = 20cc/hr, provider will assess patient for eligibility to continue to increase oxytocin dosage.
  Time frame measured from start of oxytocin infusion until the mother is discharged from hospital after giving birth.
- Obese-Intervention: 4) Intervention group: Obese cohort: BMI ≥30, at <20 weeks gestation or BMI ≥35 at a term gestation, high dose oxytocin protocol
  High dose oxytocin regimen (endorsed by American College of Obstetricians and Gynecologists): 90 units in 500cc 0.9% normal saline bag (180 milliunit/cc). Starting rate would be 6 milliunit/minute, or 2cc/hour. The medication will be increased by 6 milliunit/minute = 2cc/hr every 30 minutes until adequacy of contraction or cervical change. At 60 milliunit/minute = 20cc/hr, provider will assess patient for eligibility to continue to increase oxytocin dosage.
  Time frame measured from start of oxytocin infusion until the mother is discharged from hospital after giving birth.
Arm/Group | Lean-Control | Lean-Intervention | Obese-Control | Obese-Intervention
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/35 | 0/35 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35 | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 0/35 | 0/35 | 0/35 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-04): https://cdn.clinicaltrials.gov/large-docs/88/NCT03140488/Prot_SAP_001.pdf